CLINICAL TRIAL: NCT05327634
Title: Description of the Obstacles to Deprescribing Among French Patients Over 75 Years of Age Treated in the Geriatric Hospital Network
Brief Title: Obstacles to Deprescribing Among French Patients Over 75 Years of Age Treated in the Geriatric Hospital Network
Acronym: OUTMEDIC-FR
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD2921; 2022-A00136-37 (Other: ANSM)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-02

CONDITIONS: Medication Abuse
Keywords: Elderly patient; Inappropriate drugs; Deprescribing; Obstacles; French
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Deprescribing: Prospective study on patients aged 75 and over, hospitalised in geriatric short stay or geriatric rehabilitation units
  Interventions: Other: self-questionnaire

INTERVENTIONS:
Other: self-questionnaire — Prospective study on patients aged 75 and over, hospitalised in geriatric short stay or geriatric rehabilitation units

SUMMARY:
The aim of this study is to highlight action guidelines to encourage acceptance of deprescribing in people over 75 years of age: training, therapeutic education, post-prescription follow-up, specific patient pathways, specific consultations or even the integration of an advanced practice nurse in this process.

DETAILED DESCRIPTION:
For several years now, the proportion of senior citizens in our country has been rising steadily. There are now 6.4 million people over the age of 75 in France.

It is therefore important to take into account the needs and specificities of this part of the population. One of its particularities is polypathology. Indeed, from the age of 70 onwards, 93% of elderly subjects have at least 2 diseases and 85% have at least 3. This polypathology will lead to a large number of different prescribers with an increased risk of having more than 5 molecules in their personal treatment. This is known as polypharmacy.

In the elderly, polypharmacy is harmful. It increases the risk of adverse effects and drug interactions. In France, 20% of patients over 75 years old and 25% of those over 85 years old consult the emergency room because of adverse drug reactions.

The literature shows that we can act on these adverse events by "deprescribing". De-prescribing is defined as intentionally stopping the prescription of an unnecessary or potentially dangerous drug for a patient.

The expected benefit for the patient is to reduce the iatrogenic risks induced by treatments that would no longer be useful for him/her or that have a negative benefit/risk balance. To achieve this objective, the patient must understand this risk, understand the benefit he or she can derive from it and be an actor in this process.

For carers, the expected benefit is greater involvement of the patient in the process, better adherence to the approach, which can be organised and carried out in a safer way.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and over
* Hospitalized in geriatric short-stay or geriatric rehabilitation units
* Patients who did not object to participation in the study

Exclusion Criteria:

* Patient refusal
* Patients not able to understand and fill in the questionnaire: Cognitive disorders, Confusion, Unstable clinical state, Sensory disorders, not speaking French.
* Patient under protective supervision (guardianship or curatorship)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 and over hospitalised in geriatric short stay or geriatric rehabilitation units
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Description of the obstacles to the withdrawal of medication in patients over 75 years of age in the geriatric sector | Baseline
  The main evaluation criterion will be measured using the self-questionnaire: a revised form of the 5-point Likert-type "Revised Patients' Attitude Toward Deprescribing" (rPATD), validated in French.
  Discouragement will be assessed on the basis of the overall score of questions 1 to 20 of the self-questionnaire, with regard to questions 21 and 22.

SECONDARY OUTCOMES:
Assessment of the relationship between patient burden and acceptance (or refusal) of deprescribing. | Baseline
  They will be measured using the self-questionnaire given to patients. Responses to the burden (questions 1-5) and acceptance (question 21) questions will be measured using the revised 5-point Likert-type "Revised Patients' Attitude Toward Deprescribing" (rPATD) scale, validated in French. A correlation will be made between the two items.
  They will be measured using the self-questionnaire given to patients. Responses to the burden (questions 1-5) and acceptance (question 21) questions will be measured using the revised 5-point Likert-type "Revised Patients' Attitude Toward Deprescribing" (rPATD) scale, validated in French. A correlation will be made between the two items.
Assessment of the relationship between the benefit of the treatment experienced by the patient and the acceptance (or refusal) of the deprescribing | Baseline
  They will be measured using the self-questionnaire given to patients. Responses to the questions concerning the perceived benefit of treatment (questions 6 to 10) and acceptance (question 21) will be measured using the revised Patients' Attitude Toward Deprescribing (rPATD) 5-point Likert scale. A correlation will be made between the two items
Assessment of the relationship between concern about possible negative effects of discontinuing treatment and acceptance (or refusal) of deprescribing | Baseline
  They will be measured using the self-questionnaire given to patients. Responses to questions concerning concern about possible negative effects of stopping treatment (questions 11 to 15) and acceptance (question 21) will be measured using the revised Patients' Attitude Toward Deprescribing (rPATD) 5-point Likert scale. A correlation will be made between the two items.
Assessment of the relationship between the patient's good knowledge of their treatments and acceptance (or refusal) of the deprescribing. | Baseline
  They will be measured using the self-questionnaire given to patients. The answers to the questions concerning the patient's good knowledge of their treatments (questions 16 to 20) and acceptance (question 21) will be measured using the revised Patients' Attitude Toward Deprescribing (rPATD) 5-point Likert scale. A correlation will be made between the two items..
Assessment of the relationship between certain families of treatments and acceptance (or refusal) of deprescribing | Baseline
  They will be measured using the self-questionnaire given to patients. Responses concerning the acceptance of deprescribing according to the different treatment families will be measured using simple questions 26 to 29 of the self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Antoniazzi, Principal Investigator — Hospital René Dubos
Locations (4):
- France (4):
  - Short stay Geriatric department - Hospital Simone Veil, Beauvais
  - SSR Geriatric department - Hospital Simone Veil, Beauvais
  - Short stay Geriatric department - Hospital René Dubos, Pontoise
  - SSR Geriatric department - Hospital René Dubos, Pontoise

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roux B, Sirois C, Niquille A, Spinewine A, Ouellet N, Petein C, Sibille FX, Csajka C, Reeve E, Villeneuve C, Laroche ML. Cross-cultural adaptation and psychometric validation of the revised Patients' Attitudes Towards Deprescribing (rPATD) questionnaire in French. Res Social Adm Pharm. 2021 Aug;17(8):1453-1462. doi: 10.1016/j.sapharm.2020.11.004. Epub 2020 Nov 10. PMID 33317980
- [Derived] Antoniazzi C, Cnockaert X, Michel P. Description of barriers to the deprescription of inappropriate drugs in French hospitalized geriatric services. Sci Rep. 2025 May 15;15(1):16837. doi: 10.1038/s41598-025-99752-9. PMID 40374894